CLINICAL TRIAL: NCT06995755
Title: Atlas: An Interactive Text Messaging Program Combining Weather Alerts With Hyper-Localized Resources & Actionable Insights for Addressing Climate Change.
Brief Title: Atlas:Text Messaging Program With Weather Alerts, Local Resources & Insights for Addressing Climate Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R43ES035344 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-29 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Climate Change
MeSH Terms: interventions — POE sorbitan lanolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atlas users (Experimental): All participants were provided with access to the intervention (atlas)
  Interventions: Behavioral: atlas

INTERVENTIONS:
Behavioral: atlas — A theoretically-grounded, highly individualized text messaging intervention that 1) provided information on current climate-related and environmental risks (e.g., high temperatures, air quality alerts, asthma triggers etc.) that might adversely affect a user's current health conditions; 2) linked users to local zip-code matched resources to mitigate their specific risk (e.g., cooling centers, hurricane shelters); 3) implemented a full range of best practices in tailored health behavior change communications to personalize ongoing communications regarding the link between human actions and extreme weather based on the user's level of concern about and belief in climate change; and 4) provided customized actionable tips for addressing climate change to promote climate efficacy at the individual, community, and policy/advocacy level based on the user's level of motivation.

SUMMARY:
Climate change is an urgent public health threat, and climate-related health risks disproportionately impact vulnerable populations. To date, digital climate change communications have been limited to one-directional, one size-fits all messaging based on a single theoretical approach (i.e., framing). This Phase I SBIR explored the acceptability and effects of an innovative solution: atlas - an interactive text messaging program that leverages insights from behavior change science and integrates data from the National Weather Service to engage a broad spectrum of users with varying levels of concern about climate change and tailor the user experience.

atlas 1) provided information on current climate-related and environmental risks (e.g., high temperatures, air quality alerts, asthma triggers etc.) that might adversely affect a user's current health conditions; 2) linked users to local zip-code matched resources to mitigate their specific risk (e.g., cooling centers, hurricane shelters); 3) implemented a full range of best practices in tailored health behavior change communications to personalize ongoing communications regarding the link between human actions and extreme weather based on the user's level of concern about and belief in climate change; and 4) provided customized actionable tips for addressing climate change to promote climate efficacy at the individual, community, and policy/advocacy level based on the user's level of motivation.

Developed in collaboration with community members, 2 community health experts, and 4 climate change experts, atlas achieved sustained engagement and impact by hyper-personalizing the user experience and seamlessly integrating actionable insights from multiple theories of behavior change and communication frameworks. Extensive end user and expert input ensured atlas was designed for rapid dissemination.

Residents of a city in a New England state (n=54) were recruited to participate in a 30-day pilot test. The primary outcome, response efficacy for taking steps to mitigate climate change, was assessed across individual, collective, and governmental levels from pretest (baseline) to posttest (30-day follow-up). The hypothesis was that the atlas users will have increased response efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Being a little, moderately, very or extremely sure that climate change is happening now

Exclusion Criteria:

* Younger than 18
* Being not at all sure that climate change is happening now

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Johnson, PhD, Principal Investigator — Pro-Change Behavior Systems
Locations (1):
- Pro-Change Behavior Systems, Narragansett, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
A variety of peer-reviewed publications will emerge from the proposed research. At the conclusion of the study, the data will be de-identified and then made available to those requesting access, provided that they sign an agreement that the data will be used for research purposes only. Pro-Change routinely asks those requesting access to any data to sign such a form.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atlas Users
Started | 54
Completed | 46
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Atlas Users
Number analyzed (Participants) | 54
Age, Customized [Mean (Standard Deviation); unit: years] | 42.2 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 21
  Hispanic | 12
  Other | 12
  White | 9
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Response Efficacy Scale
Description: A 3-item measure of response efficacy that assessed individual, community, and governmental/policy level efficacy for mitigating climate change. It is measured using a Likert scale, with total scores ranging from 3 to 15. Higher scores reflect a better outcome.
Time Frame: Pretest (baseline) and Posttest (30 day follow-up)
Population: 36 users completed baseline & follow-up and did not have a maximum score on response efficacy measure (a score of 15), in which case they were excluded from the primary outcome analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atlas Users
Number analyzed (Participants) | 36
score on a scale
  Pretest (baseline) | 9.69 (2.87)
  Posttest (30 day follow-up) | 10.86 (2.64)

2. Secondary Outcome: Confidence
Description: This 3-item scale assesses an individual's confidence level in taking at least one climate friendly action in the next month. Ratings of confidence will be made on a 5-point Likert scale (1=not at all; 5=extremely confident). Raw scores range from a minimum of 3 to a maximum of 15, with higher scores indicating better outcomes.
Time Frame: Pretest (baseline) and Posttest (30 day follow-up)
Population: 16 of the 46 users reported max scores in confidence thus were not included in outcome analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atlas Users
Number analyzed (Participants) | 30
score on a scale
  Pretest (baseline) | 3.03 (0.85)
  Posttest (30 day follow-up) | 3.70 (1.12)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 30 days
Arm/Group | Atlas Users
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT06995755/Prot_003.pdf
  • Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT06995755/SAP_004.pdf
  • Informed Consent Form (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT06995755/ICF_005.pdf